CLINICAL TRIAL: NCT02261584
Title: Comparative Study of Microwave Ablation and Partial Splenic Embolization in the Management of Hypersplenism
Brief Title: Microwave Ablation and Partial Splenic Embolization in the Management of Hypersplenism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Shebl, Dr., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microwave vs PSE
Record Dates: First submitted 2014-09-26; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Hypersplenism
MeSH Terms: conditions — Hypersplenism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Microwave Thermal Coagulation (Experimental): MW ablation performed either laparoscopically or percutaneously is a safe, effective, and minimally invasive technique for the management of hypersplenism in patients with liver cirrhosis. It may significantly increase platelet count and white blood cell (WBC) count and improve hepatic blood supply with fewer complications. Ablating more than 40% of the splenic parenchyma may yield better long term results. This method may provide a new and promising minimally invasive alternative for treating hypersplenism.
  Interventions: Device: Microwave Thermal Coagulation
- Partial Splenic Embolization Catheter (Experimental): Partial splenic embolization (PSE), which was first performed by Spigos et al in 1979, has been considered first-line therapy for hypersplenism in many institutions, and has been proposed as an effective alternative to splenectomy for improving peripheral blood cell counts. However, PSE is associated with many complications, including intermittent fever, abdominal pain, nausea, vomiting, post-embolization syndrome, splenic abscess, splenic rupture, pneumonia, refractory ascites, pleural effusion and gastrointestinal bleeding. To ensure a sustained and long-term increase in platelet and leucocytic counts, the splenic infarction rate needs to be greater than 50% (8). Thus, severe complications can ensue.
  Interventions: Device: Partial Splenic Embolization

INTERVENTIONS:
Device: Microwave Thermal Coagulation — Microwave thermal coagulation of splenic parenchyma.
  Other Names: Microwave
  Arms: Microwave Thermal Coagulation
Device: Partial Splenic Embolization — Femoral artery approach will be used for splenic artery catheterization with the tip of the catheter always well advanced selectively into the splenic artery. Embolizing agent will be injected in small increments. Arteriography in between divided doses will be done to document the extent of devascularization.
  Other Names: PSE
  Arms: Partial Splenic Embolization Catheter

SUMMARY:
The aim of this study is to compare microwave thermal coagulation and partial splenic embolization in the management of hypersplenism in patients with cirrhosis.

This study will be conducted on 40 patients with liver cirrhosis associated with splenomegaly and hypersplenism. The study will be done at the National Hepatology and Tropical Medicine Research Institute.

DETAILED DESCRIPTION:
Liver cirrhosis or portal hypertension is frequently associated with congestive splenomegaly resulting in hypersplenism.

Hypersplenism can be defined as anemia, leukopenia, thrombocytopenia, or a combination of these resulting from excessive, splenic sequestration or pooling of blood cells, usually associated with clinical splenomegaly and always ameliorated by splenectomy.

Partial splenic embolization (PSE), which was first performed by Spigos et al in 1979, has been considered first-line therapy for hypersplenism in many institutions, and has been proposed as an effective alternative to splenectomy for improving peripheral blood cell counts. However, PSE is associated with many complications, including intermittent fever, abdominal pain, nausea, vomiting, post-embolization syndrome, splenic abscess, splenic rupture, pneumonia, refractory ascites, pleural effusion and gastrointestinal bleeding. To ensure a sustained and long-term increase in platelet and leucocytic counts, the splenic infarction rate needs to be greater than 50%. Thus, severe complications can ensue.

Thermal ablation methods using different energy sources, such as radiofrequency (RF), microwave (MW), or laser, were developed rapidly as minimally invasive techniques for the eradication of local tumor tissue within solid organs. There have been reports of the use of radiofrequency to ablate normal spleen, splenic injury, and splenomegaly.

Radiofrequency Ablation (RFA) had comparable efficacy and a better safety than PSE in the treatment of hypersplenism in patients with post hepatitis c cirrhosis.

MW ablation performed either laparoscopically or percutaneously is a safe, effective, and minimally invasive technique for the management of hypersplenism in patients with liver cirrhosis. It may significantly increase platelet count and white blood cells (WBC) count and improve hepatic blood supply with fewer complications. Ablating more than 40% of the splenic parenchyma may yield better long term results. This method may provide a new and promising minimally invasive alternative for treating hypersplenism.

The aim of this study is to compare microwave thermal coagulation and partial splenic embolization in the management of hypersplenism in patients with cirrhosis.

This study will be conducted on 40 patients with liver cirrhosis associated with splenomegaly and hypersplenism. The study will be done at the National Hepatology and Tropical Medicine Research Institute.

All patients will be subjected to thorough history taking, full clinical, lab, ultrasound/doppler, and upper endoscopic examination. Diagnosis has been based on peripheral blood count and confirmed with bone marrow examination.

Preoperative antibiotics will be given and correction of bleeding tendency with plasma and platelet transfusion will be done as required to get a prothrombin concentration more than 65% and platelet count more than 100,000.

ELIGIBILITY:
Inclusion Criteria:

* Liver Cirrhosis
* Hypersplenism

Exclusion Criteria:

* Patients with bad performance scale.
* Patients with hepatic encephalopathy and tense ascites.
* Patient with active esophageal variceal bleeding .
* Patients with hypocellular bone marrow (BM).
* Patients with renal failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with improvement of hypersplenism after microwave thermal coagulation of the spleen compared with partial splenic embolization. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, MD, Principal Investigator — Tanta Faculty of Medicine, Professor; Fat-heya E Assel, MD', Study Director — Tanta Faculty of Medicine, Professor; Mohamed M Elkassas, Study Director — Dr.; Islam S Ismail, Study Director — Dr.
Locations (1):
- National Hepatology and Tropical Medicine Research Institute, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Result] Pursnani KG, Sillin LF, Kaplan DS. Effect of transjugular intrahepatic portosystemic shunt on secondary hypersplenism. Am J Surg. 1997 Mar;173(3):169-73. doi: 10.1016/s0002-9610(97)00006-8. PMID 9124620
- [Result] Spigos DG, Jonasson O, Mozes M, Capek V. Partial splenic embolization in the treatment of hypersplenism. AJR Am J Roentgenol. 1979 May;132(5):777-82. doi: 10.2214/ajr.132.5.777. PMID 107745
- [Result] Tajiri T, Onda M, Yoshida H, Mamada Y, Taniai N, Kumazaki T. Long-term hematological and biochemical effects of partial splenic embolization in hepatic cirrhosis. Hepatogastroenterology. 2002 Sep-Oct;49(47):1445-8. PMID 12239963
- [Result] Sangro B, Bilbao I, Herrero I, Corella C, Longo J, Beloqui O, Ruiz J, Zozaya JM, Quiroga J, Prieto J. Partial splenic embolization for the treatment of hypersplenism in cirrhosis. Hepatology. 1993 Aug;18(2):309-14. PMID 8340060
- [Result] N'Kontchou G, Seror O, Bourcier V, Mohand D, Ajavon Y, Castera L, Grando-Lemaire V, Ganne-Carrie N, Sellier N, Trinchet JC, Beaugrand M. Partial splenic embolization in patients with cirrhosis: efficacy, tolerance and long-term outcome in 32 patients. Eur J Gastroenterol Hepatol. 2005 Feb;17(2):179-84. doi: 10.1097/00042737-200502000-00008. PMID 15674095
- [Result] Hayashi H, Beppu T, Okabe K, Masuda T, Okabe H, Baba H. Risk factors for complications after partial splenic embolization for liver cirrhosis. Br J Surg. 2008 Jun;95(6):744-50. doi: 10.1002/bjs.6081. PMID 18412294
- [Result] Zhu K, Meng X, Qian J, Huang M, Li Z, Guan S, Jiang Z, Shan H. Partial splenic embolization for hypersplenism in cirrhosis: a long-term outcome in 62 patients. Dig Liver Dis. 2009 Jun;41(6):411-6. doi: 10.1016/j.dld.2008.10.005. Epub 2008 Dec 12. PMID 19070555
- [Result] Matsuoka T, Yamamoto A, Okuma T, Oyama Y, Nakamura K, Inoue Y. CT-guided percutaneous radiofrequency ablation of spleen: a preliminary study. AJR Am J Roentgenol. 2007 Apr;188(4):1044-6. doi: 10.2214/AJR.06.0641. PMID 17377043
- [Result] Felekouras E, Kontos M, Pissanou T, Pikoulis E, Drakos E, Papalambros E, Diamantis T, Bastounis E. A new spleen-preserving technique using radiofrequency ablation technology. J Trauma. 2004 Dec;57(6):1225-9. doi: 10.1097/01.ta.0000145072.31725.52. PMID 15625453
- [Result] Liu Q, Ma K, He Z, Dong J, Hua X, Huang X, Qiao L. Radiofrequency ablation for hypersplenism in patients with liver cirrhosis: a pilot study. J Gastrointest Surg. 2005 May-Jun;9(5):648-57. doi: 10.1016/j.gassur.2004.11.006. PMID 15862259
- [Result] Wasfi et al., Prospective randomized controlled study of Radiofrequency Ablation and Partial Splenic Embolization in the Treatment of Hypersplenism in patients with post-hepatitis C cirrhosis. AASLD poster DDW 2014, Chicago, USA
- [Result] Liang P, Gao Y, Zhang H, Yu X, Wang Y, Duan Y, Shi W. Microwave ablation in the spleen for treatment of secondary hypersplenism: a preliminary study. AJR Am J Roentgenol. 2011 Mar;196(3):692-6. doi: 10.2214/AJR.10.4193. PMID 21343515
- [Result] Rasekhi AR, Naderifar M, Bagheri MH, Shahriari M, Foroutan H, Karimi M, Nabavizadeh SA. Radiofrequency ablation of the spleen in patients with thalassemia intermedia: a pilot study. AJR Am J Roentgenol. 2009 May;192(5):1425-9. doi: 10.2214/AJR.08.1382. PMID 19380572
- [Result] Crooks V, Waller S, Smith T, Hahn TJ. The use of the Karnofsky Performance Scale in determining outcomes and risk in geriatric outpatients. J Gerontol. 1991 Jul;46(4):M139-44. doi: 10.1093/geronj/46.4.m139. PMID 2071835